CLINICAL TRIAL: NCT06288256
Title: Neurocognitive and Genomic Predictors of Persistent Pain and Opioid Misuse After Spine Surgery
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Chinwe Nwaneshiudu, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-22-01390
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Spine Pathology; Elective Spine Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults Undergoing Spine Surgery: Adults Undergoing Spine Surgery on opiods
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Having spine surgery and recovery is a vulnerable period when opioid naive patients may transition into long-term use of opioids, and when previously opioid tolerant patients may be at risk to continue towards long-term opioid use and dependence. However, little is known about risk for developing opioid misuse, taking opioids differently than indicated or prescribed, and later OUD. This study addresses the question of whether behavior, cognitive features, and genomic markers can predict misuse of opioids, persistent pain and disability in individuals after spine surgery.

To determine if impulsivity, inhibitory control, drug choice, and/or cognitive distortions predict opioid misuse and disability in spine surgery patients with differential gene expression.

This is a prospective observational longitudinal study characterizing behavioral phenotypes in adults undergoing spine surgery using both patient-reported survey measures, cognitive testing and blood sampling. Outcome measures include correlations between impulsivity measures, opioid drug choice responses and cognitive distortion scores, and opioid misuse with spine related disability, and gene expression counts.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* With diagnoses of lumbar, cervical or thoracic spine pathology, scheduled to undergo elective spine surgery with or without instrumentation

Exclusion Criteria:

* Severe psychiatric condition interfering with study participation Any major cardiac, pulmonary, renal, infectious, hepatic condition that interferes with study participation
* Polytrauma
* Prolonged hospitalization (>10days)
* Pregnancy
* Known surgery cancellation within study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: undergoing elective spine surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Current Opioid Misuse Measure (COMM) Score | Up to 12 months post-operatively
  The Current Opioid Misuse Measure (COMM) is a 17-item self-report measure with total scores ranging from 0 to 68 that is used to identify risk of opioid misuse among chronic pain patients, with higher scores indicating higher risk of opioid misuse.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) Score | Up to 12 months post-operatively
  The Numerical Rating Scale (NRS) for pain intensity is an 11-point scale ranging from 0 to 10 that is used to measure a patient's self-reported pain intensity, with higher scores indicating more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Chinwe Nwaneshiudu, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Spine Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis.
  Proposals should be directed to chinwe.nwaneshiudu@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third-party website (TBD).